CLINICAL TRIAL: NCT02271009
Title: A Double-Blind, Placebo-Controlled, Randomized Trial to Compare the Efficacy and Tolerability of Three Dose Regimens of AllerT, in Adults With Allergic Rhino-Conjunctivitis to Birch Pollen Studied in Environmental Exposure Chamber
Brief Title: Compare Dose Regimens of AllerT, in Adults With Allergic Rhino-Conjunctivitis to Birch Pollen Studied in EEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anergis (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN008T
Record Dates: First submitted 2014-10-14; First posted 2014-10-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Allergic Rhino-Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo without Al(OH)3 (Placebo Comparator): Five (5) SC injections over a two-month (8-week) period, according to the following schedule:
  * First three SC injections at weekly intervals.
  * Fourth SC injection two weeks after the third injection.
  * Fifth SC injection four weeks after the fourth injection.
  Interventions: Drug: Placebo
- AllerT (10 µg with Al(OH)3) (Active Comparator): Five (5) SC injections over a two-month (8-week) period, according to the following schedule:
  * First three SC injections at weekly intervals.
  * Fourth SC injection two weeks after the third injection.
  * Fifth SC injection four weeks after the fourth injection.
  Interventions: Drug: AllerT
- AllerT (25 µg with Al(OH)3) (Active Comparator): Five (5) SC injections over a two-month (8-week) period, according to the following schedule:
  * First three SC injections at weekly intervals.
  * Fourth SC injection two weeks after the third injection.
  * Fifth SC injection four weeks after the fourth injection.
  Interventions: Drug: AllerT
- AllerT (50 µg with Al(OH)3) (Active Comparator): Five (5) SC injections over a two-month (8-week) period, according to the following schedule:
  * First three SC injections at weekly intervals.
  * Fourth SC injection two weeks after the third injection.
  * Fifth SC injection four weeks after the fourth injection.
  Interventions: Drug: AllerT

INTERVENTIONS:
Drug: AllerT — Ultrafast immunotherapy
  Other Names: Continuous overlapping peptides
  Arms: AllerT (10 µg with Al(OH)3); AllerT (25 µg with Al(OH)3); AllerT (50 µg with Al(OH)3)
Drug: Placebo — placebo control
  Arms: Placebo without Al(OH)3

SUMMARY:
The purpose of this study is to find the optimal dose of AllerT that should be used to treat moderate to severe allergies due to birch tree pollen.

There are 4 treatment groups in this study; 3 treatment groups will receive AllerT at different doses and 1 treatment group will receive placebo.

This study will also assess the effectiveness and safety of AllerT compared to placebo in relieving allergy symptoms.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the dose-response trend of three doses of adjuvanted AllerT and of placebo in reducing symptoms of allergic rhino-conjunctivitis in subjects exposed to birch tree pollen in an environmental exposure chamber (EEC).

Secondary Objectives:

* To evaluate three dose regimens of AllerT , versus a placebo in reducing symptoms of allergic rhino-conjunctivitis in subjects exposed to birch tree pollen in an EEC.
* To assess the safety and tolerability of a two month treatment with three dose regiments of AllerT (10 µg, 25 µg and 50 µg with Al(OH)3).
* To explore the immunological response to AllerT.

ELIGIBILITY:
Inclusion Criteria:

* Minimum two-year history of moderate to severe rhino-conjunctivitis on exposure to birch pollen with a need to take symptomatic medications (antihistamine, steroid) during pollen season, prior to study enrollment.
* Sensitivity to birch tree pollen confirmed at Screening by both of the following criteria:
* Positive Skin Prick Test (SPT) to birch pollen extract (wheal ≥ 3 mm than the negative control). Negative control must be ≤ 2 mm.
* Positive specific IgE CAP test for Bet v 1 (≥ 0.7 kU/L).
* A qualifying score in at least one of the two Baseline EEC Challenges: at least one diary card of 12/24 or greater for Total Rhinoconjunctivitis Symptom Score (TRSS) as well as either one diary card 6/12 or greater for Total Nasal Symptom Score (TNSS) or Total Ocular Symptom Score (TOSS).

Exclusion Criteria:

* Positive SPT to AllerT (wheal ≥ 3 mm than the negative control).
* Received specific immunotherapy against:

  * Any allergen within three years before the Screening visit.
  * Birch tree pollen or a tree pollen mix including birch pollen at any time before the Screening visit.
* Clinically significant symptoms due to allergens other than birch pollen during the EEC challenge periods (eg, perennial allergies, allergies to other pollens with overlapping allergy seasons during the EEC periods).
* Persistent un-controlled asthma; subjects with a Forced Expiratory Volume (FEV1) lower than 80% of their predicted value and/or subjects under chronic treatment for asthma with regular use of inhaled steroids. Subjects with seasonal asthma may be included. Subjects who require the occasional use of inhaled broncho-dilator can be included.
* History of birch pollen induced asthma. Note: A diagnosis of isolated exercise induced bronchospasm or controlled asthma (Global Initiative for Asthma [GINA] Step 1) not triggered by birch pollen does not constitute an exclusion criterion.
* History of documented severe anaphylactic reaction (Grade 4 of World Allergy Organization [WAO]).
* History of sinus disease including:

  * Acute or significant chronic sinusitis.
  * History of significant recurrent acute sinusitis, defined as two episodes per year for the last two years, all of which required antibiotic treatment.
  * History of chronic sinusitis, defined as sinus symptoms lasting greater than 12 weeks that includes two or more major factors or one major factor and two minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, and ear pain, pressure, or fullness.
* Subjects who cannot tolerate the Baseline EEC Challenge or do not meet the Baseline EEC Challenge inclusion criteria.
* Subjects with a history of immunodeficiency or any other conditions that might affect the subject's safety or interpretation of study results.
* Received immunosuppressive medication (including oral corticosteroids) within four weeks prior to Screening, or planned to be used during the trial period.
* Received systemic or local antihistamines, oral or inhaled corticosteroids or under antidepressant medication with antihistamine effects within two weeks prior to Screening.
* Subjects for whom administration of epinephrine is contraindicated (eg, subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* Subjects being treated with beta-blockers in any form including topical ocular beta-blocker type medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The change in average Total Rhinoconjunctivitis Symptom Scores (TRSS) from the Baseline EEC Challenge (Visit 1 & Visit 2) to the Post-Treatment EEC Challenge (PTC) (Visit 8 & Visit 9). | before entry in the EEC (time point = 0) and then every 30 minutes up to 6 hours in the EEC (12 time points)
  The mean TRSS will be calculated for each subject from t =1 hour to t = 6 hours inclusive for the 2 consecutive days (22 time points) of Baseline and post-treatment EEC challenge.

SECONDARY OUTCOMES:
Individual Nasal Symptom Scores (NSS) | from t =1 hour to t = 6 hours inclusive for the 2 consecutive days (22 time points) of Baseline and post-treatment EEC challenge
  • The change in the average of individual NSS from the Baseline EEC Challenge (Visit 1 & Visit 2) to the Post-Treatment EEC Challenge (Visit 8 & Visit 9).
Individual NSS | All time points in the EEC for the 2 consecutive days (24 time points) of Baseline and post-treatment EEC challenge
  Individual NSS from Baseline EEC Challenge (Visit 1 & Visit 2) to Post-Treatment EEC Challenge (Visit 8 & Visit 9) (24 time points).
The Global Evaluation of Treatment Efficacy Questionnaire | Visit 9, after the last post-treatment EEC session.
The Asthma Symptom Score (ASS) | before entry in the EEC (time point =0) and then every 30 minutes up to 6 hours in the EEC (12 time points)
  The mean ASS will be calculated for each subject from t =1 hour to t = 6 hours inclusive for the 2 consecutive days of the EEC challenge (22 time points). The following will be analyzed:
  * The change in the average ASS from the Baseline EEC Challenge (Visit 1 & Visit 2) to the Post-Treatment EEC Challenge (Visit 8 & Visit 9).
  * The change in the pre-EEC-Specific Quality of Life Questionnaire (EEC-Specific QoLQ) to post EEC-QoLQ will be calculated at Baseline EEC Challenge (Visit 1 & Visit 2) and at Post-Treatment EEC Challenge (PTC) (Visit 8 & Visit 9). Change of (post- pre-EEC) form Baseline to PTC will be compared between treatment groups.
The mean TRSS | All time points in the EEC for the 2 consecutive days (24 time points) of Baseline and post-treatment EEC challenge
  The following will be analyzed:
  * The change in the average TRSS, from Baseline EEC Challenge (Visit 1 & Visit 2) to Post-Treatment EEC Challenge (Visit 8 & Visit 9) (24 time points).
  * The change in the average TRSS from the Baseline EEC Challenge (Visit 1, 12 time points) to the Post-Treatment EEC Challenge (Visit 8, 12 time points) will be calculated.
The mean TNSS | All time points in the EEC for the 2 consecutive days (24 time points) of Baseline and post-treatment EEC challenge
  The following will be analyzed:
  * The change in the average TNSS from Baseline EEC Challenge (Visit 1 & Visit 2) to Post-Treatment EEC Challenge (Visit 8 & Visit 9) (24 time points).
  * The change in the average TNSS from the Baseline EEC Challenge (Visit 1, 12 time points) to the Post-Treatment EEC Challenge (Visit 8, 12 time points) will be calculated.
The mean TOSS | All time points in the EEC for the 2 consecutive days (24 time points) of Baseline and post-treatment EEC challenge
  The following will be analyzed:
  * The change in the average TOSS from Baseline EEC Challenge (Visit 1 & Visit 2) to Post-Treatment EEC Challenge (Visit 8 & Visit 9) (24 time points).
  * The change in the average TOSS from the Baseline EEC Challenge (Visit 1, 12 time points) to the Post-Treatment EEC Challenge (Visit 8, 12 time points) will be calculated.
The mean Total Nasal Symptom Scores (TNSS) | from t =1 hour to t = 6 hours inclusive for the 2 consecutive days (22 time points) of Baseline and post-treatment EEC challenge
  The following will be analyzed:
  • The change in the average TNSS from the Baseline EEC Challenge (Visit 1 & Visit 2) to the Post-Treatment EEC Challenge (Visit 8 & Visit 9).
Total Ocular Symptom Score (TOSS) | before entry in the EEC (time point = 0) and then every 30 minutes up to 6 hours in the EEC (12 time points)
  • The changes in the average TOSS from the Baseline EEC Challenge (Visit 1 & Visit 2) to the Post-Treatment EEC Challenge (Visit 8 & Visit 9).

OTHER OUTCOMES:
The change in Bet v 1 specific immunoglobulin (Ig)E and IgG4 and AllerT specific IgE and IgG4. | Screening Day 166 upto Day 3, Day 0
The change in Bet v 1 specific immunoglobulin (Ig)E and IgG4 and AllerT specific IgE and IgG4. | Day 0, Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada